CLINICAL TRIAL: NCT01441323
Title: USC Center for Transdisciplinary Research on Energetics and Cancer or Obesity-Related Metabolic Disease Risk: Response to Exercise in Minority Youth
Brief Title: Strength Training and Nutrition Development for African American Youth
Acronym: STAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael I. Goran, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 195-1642394A1; 1U54CA116848 (NIH)
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Obesity; Type 2 Diabetes; Cardiovascular Risk; Cancer
Keywords: Obesity; Type 2 Diabetes; Cardiovascular Risk; Cancer; African American; Adolescents; Strength Training; Nutrition
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Neoplasms | interventions — Nutritional Status; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (C) (No Intervention)
- Nutrition (N) (Experimental)
  Interventions: Behavioral: Nutrition
- Strength Training & Nutrition (ST) (Experimental)
  Interventions: Behavioral: Strength Training & Nutrition

INTERVENTIONS:
Behavioral: Nutrition — Nutrition classes for 1 hour & 30 minutes once a week for 16 weeks + motivational interviewing (4 individual sessions)
  Arms: Nutrition (N)
Behavioral: Strength Training & Nutrition — Strength Training twice a week for 1 hour a day for 16 weeks + Nutrition once a week for 1 hour & 30 minutes for 16 weeks + motivational interviewing (4 individual & 4 group sessions)
  Arms: Strength Training & Nutrition (ST)

SUMMARY:
The investigators are conducting an intervention study to examine the effects of a 16-week exercise and diet interventions on prevention of disease, specifically type 2 diabetes and heart disease, in African American youth. Sixty overweight African American boys and girls will be recruited and placed in one of the following intervention groups: 1) Control Group (delayed intervention), 2) Dietary Education Group (nutrition education focused on reducing sugar & soda, increased fiber & whole grain intake), or 3) Combination of Strength Training (twice/week for 60 min, progressive increases in exercise volume and intensity) + Dietary Education (nutrition education focused on reducing sugar & soda, increased fiber & whole grain intake). The investigators will assess which intervention group has the most effects on health parameters such as weight, body composition, and insulin related measures.

DETAILED DESCRIPTION:
A.1 Aims

The overall goal of this project is to examine role of strength training as a therapeutic intervention to improve the cancer and obesity-related metabolic risk profile in African-American adolescents. The project is prompted by the urgent public health need to prevent and treat cancer and obesity-related problems, including diabetes and cardiovascular disease, in African-American adolescents, a population that is understudied and medically under-served in the Los Angeles area. A recent report from the Institute of Medicine underscored this major public health concern in the childhood obesity field:

"Children's health has made tremendous strides over the past century. In general, life expectancy has increased by more than thirty years since 1900 and much of this improvement is due to the reduction of infant and early childhood mortality. Given this trajectory toward a healthier childhood, the investigators begin the 21st century with a shocking development - an epidemic of obesity in children and youth. The increased number of obese children throughout the US during the past 25 years has led policymakers to rank it as one of the most critical public health threats of the 21st century. (92)" Obesity and metabolic syndrome problems disproportionately affect African-American adolescents (51). This project will explore why African-Americans have greater cancer risk than Hispanics (91), despite a reduced prevalence of the metabolic syndrome (7, 62).

Preliminary work from this laboratory has shown that both African-American and Hispanic children are more insulin resistant than Caucasian children, and this difference is apparently not explained by differences in body fatness. Moreover, the metabolic compensation to a similar degree of insulin resistance markedly differs between African-American and Hispanic children (62). African-Americans display greater hyperinsulinemia in response to a glucose challenge, whereas Hispanics have a more subdued increase in insulin levels due to an increase in second phase insulin secretion. The investigators will have the opportunity to build upon this preliminary work to examine the effects of resistance training on three factors predictive of cancer and metabolic disease risk: 1) body fat distribution; 2) insulin resistance and 3) measures of oxidative stress in African America adolescents. The investigators previously studying Hispanic adolescents in a parallel protocol.

The overall hypotheses of this project are that: (1) hyperinsulinemia in overweight African-American youth is associated with increased long-term cancer risk; and (2) insulin resistance, obesity and oxidative stress in overweight African-American youth will be improved with chronic resistance training and a modified carbohydrate dietary approach. The investigators will specifically examine the following metabolic outcomes, because they have been hypothesized to contribute to the obesity-related increase in cancer and metabolic disease risk:

* Insulin concentrations and insulin sensitivity;
* Total body fat, abdominal visceral fat, muscle fat and liver fat;
* Circulating adipocytokines;
* Intima-media thickness of the carotid artery
* Markers of oxidative stress, including: F2-isoprostanes, malondialdehyde (MDA), myeloperoxidase (MPO), oxygen radical absorbance capacity and ROS detection by flow cytometry.

A.2 Aims

The specific aims and hypotheses of project 1 are as follows:

Study 1: Cross-Sectional Measures Specific Aim 1 (Body Fat Compartments): To determine the association of visceral fat, muscle and liver fat and plasma adipocytokines to variation in insulin resistance in African-American youth.

* Hypothesis 1: Visceral fat, muscle and liver fat, and adipokines will independently contribute to greater insulin resistance.

  • Specific Aim 2 (Insulin Resistance): To examine metabolic compensation to insulin resistance in African-American youth.
* Hypothesis 2: Insulin resistant African-American youth will exhibit a higher acute insulin response to glucose.

  • Specific Aim 3 (Oxidative Stress): To examine the influence of body fat and insulin resistance on markers of oxidative stress and markers of metabolic disease risk.
* Hypothesis 3: Increased total body fat and insulin resistance will be associated with greater oxidative stress. The increased oxidative stress will be correlated with the higher acute insulin response.

Study 2 (Randomized Trial of Modification of Carbohydrate Intake and Strength Training) • Specific Aim 4 (Linkage of factors in Aims 1-3): To determine the effects of a randomized modification of carbohydrate intake, and/or strength training intervention in overweight African-American adolescents on potential factors linking obesity, insulin resistance, and oxidative stress.

- Hypothesis 4: Strength training will improve metabolic factors for cancer risk. That is, resistance training will reduce visceral fat; increase insulin sensitivity, reduce hyperinsulinemia, and reduce oxidative stress. The decreases in total body fat and visceral adipose tissue will be associated with improved insulin sensitivity and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (≥85th BMI percentile)
* African American: Children will initially be defined as African American if they and both parents and all 4 grandparents self identify as African American.

Exclusion Criteria:

* Diabetes: Children will not be eligible for participation if they have any diagnostic criteria for diabetes, including polyuria, polydipsia with or without unexplained weight loss, fasting plasma glucose >126 mg/dl, or a 2-hour plasma glucose >200 mg/dL during an OGTT using a dose of 1.75g glucose/kg BW (to a maximum of 75g). Children will also be excluded if they test positive for diabetes-related auto-antibodies, including ICA512 and GAD. Children testing positive for type 2 diabetes will be referred for treatment. Children with impaired glucose tolerance (fasting glucose >100 mg/dL or 2-hour glucose >140 mg/dl during an oral glucose tolerance test) and/or conditions associated with insulin resistance (e.g. acanthosis nigricans, hypertension, dyslipidemia, poly-cystic ovarian syndrome) will be eligible, as long as they are not receiving treatment and meet other eligibility criteria.
* Weight loss or exercise program: currently involved with any weight loss or exercise program, or have been in the 6 months prior to participation
* Use of medications: taking any medications known to influence body composition or insulin action/secretion (e.g. prednisone, ritalin, growth hormone)
* Syndromes that influence body composition: diagnosed with syndromes or diseases that may influence body composition and fat distribution (e.g. Cushing syndrome, Down syndrome)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | post interventive (week 16)

SECONDARY OUTCOMES:
adiposity | post intervention (week 16)

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, PhD, Principal Investigator — University of Southern California
Locations (1):
- Veronica Atkins Lifestyle Intervention Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hijazin K, Smith B, Garrett C, Knox A, Kelly LA. Relationship between adiponectin and blood pressure in obese Latino adolescent boys with a family history of type 2 diabetes. BMC Pediatr. 2023 Oct 20;23(1):523. doi: 10.1186/s12887-023-04337-y. PMID 37864156